CLINICAL TRIAL: NCT04886505
Title: An Early Feasibility Study Assessing the Safety, Technical Performance, and Efficacy of the Electrolytic eCLIPs Bifurcation System for the Treatment of Intracranial Bifurcation Aneurysms
Brief Title: An EFS Assessing the Electrolytic eCLIPs System for Treatment of Intracranial Aneurysms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds
Sponsor: Evasc Medical Systems Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS 20-018
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2021-09

CONDITIONS: Aneurysm, Intracranial
Keywords: Bifurcation aneurysm; Coil retention; Flow diversion
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Single arm study - treatment with Electrolytic eCLIPs Bifurcation System
  Interventions: Device: Electrolytic eCLIPs Bifurcation System

INTERVENTIONS:
Device: Electrolytic eCLIPs Bifurcation System — The electrolytic eCLIPs bifurcation system will be implanted into patients with bifurcated saccular intra-cranial aneurysms.

SUMMARY:
The purpose of this study is to investigate the feasibility and initial clinical safety of eCLIPs device use for the treatment of wide-necked bifurcation aneurysms. The eCLIPs device is a novel shield like implant that is placed across the neck of the aneurysm and not only facilitates coil retention but also partly obstructs the flow of blood into the aneurysm.

This is an early feasibility study, which is a small study investigating an innovative device to gather more clinical data before conducting a larger study. The safety and the effects of the device on the aneurysm will be studied for 12 months after the procedure among 15 patients at approximately 4 participating hospital centers. A larger study will be required to determine the safety and efficacy of the eCLIPs device for the treatment of wide-necked bifurcation aneurysms.

DETAILED DESCRIPTION:
The primary objective of this study is to obtain preliminary confirmation that the eCLIPs Delivery Wire is safe and provides sufficient technical performance in delivering the eCLIPs Implant to distal tortuous anatomies.

This study will be a multicentre, open label, single-arm safety, technical performance, and efficacy study of the Electrolytic eCLIPs Bifurcation System in the management of bifurcated intracranial aneurysms (IA). Subjects included in the study will have saccular intracranial aneurysms that arise at or adjacent to a bifurcation, having a neck length of ≥ 4mm or have a dome:neck ratio <2. Aside from the implantation of the eCLIPs Implant, the study will follow usual clinical care practices.

The subjects will undergo clinical assessments at pre-discharge and 30 days, as well as clinical assessment and radiographic imaging at 6 and 12 months (Digital Subtraction Angiography; DSA).

It is important to note that changes to the investigational device may occur during the course of this early feasibility study. Ongoing results of the study will be evaluated, along with collection of detailed operator feedback on usability, in order to determine whether further refinements to the eCLIPs Delivery Wire are required.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with an unruptured or previously ruptured (at least 1 month from date of rupture and with partial occlusion of the dome of the aneurysm by endovascular techniques or by open neurosurgery, and in stable neurological condition-WFNS I and II with a good recovery to at least to mRS 0-2) saccular, intracranial aneurysm or recurrent aneurysm with maximal diameter <25mm and has a neck length of > 4mm or dome:neck ratio <2, arising at a bifurcation with branch artery diameters of 1.5mm to 3.25mm:
2. Patient understands the nature of the procedure and has the capacity to provide informed consent.
3. Patient is willing to have on-site follow-up evaluations up to 5-yrs
4. In the clinician's judgement, the aneurysm requires intervention, given risk of rupture or other rationale (as documented on the Screening CRF), and that the patient agrees with that clinician judgement

Exclusion Criteria:

1. Patient who presents with an intracranial mass or currently undergoing radiation therapy for carcinoma of the head or neck region.
2. Major surgery within previous 30 days or planned within 120 days after enrolment.
3. Patient with an International Normalized Ratio (INR)≥ 1.5.
4. Patient with serum creatinine level ≥104 μmol/L (or 2.5mg/dL) at time of enrolment.
5. Patient with a platelet count ˂100x103 cells/mm3 or known platelet dysfunction at time of enrolment
6. Patient who has a known cardiac disorder, likely to be associated with cardioembolic symptoms such as atrial fibrillation
7. Patient with any condition that, in the opinion of the treating physician, would place the subject at a high risk of embolic stroke or with any medical co-morbidity likely to affect the outcome (e.g. pulmonary disease, uncontrolled diabetes, blood disorders).
8. Patient with known allergies to nickel-titanium metal
9. Patient with known allergies to aspirin, heparin, ticlopidine, clopidogrel, prasugrel or other anti-platelet or P2Y12 agents or to general anesthesia.
10. Patient with resistance to P2Y12 agents based on a validated platelet testing method (Verify Now, Multiplate or other).
11. Patient with a life-threatening allergy to contrast (patients with itching or rash as a reaction to contrast can be included if properly prophylactically treated).
12. Patient with inappropriate anatomy as demonstrated by angiography due to severe intracranial vessel tortuosity or stenosis, or intracranial vasospasm not responsive to medical therapy.
13. Patient who is currently participating in another clinical research study involving an investigational product.
14. Patient who has had a previous intracranial procedure associated with the target aneurysm such that access and placement of an eCLIPS device would be compromised
15. Stenting, angioplasty, or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to the treatment date.
16. More than one intracranial aneurysm that requires treatment within 12 months.
17. Asymptomatic extradural aneurysms requiring treatment.
18. Severe neurological deficit that renders the patient incapable of living independently.
19. Unstable neurological deficit (i.e. worsening or improvement of clinical condition in the last 30 days.
20. Dementia or psychiatric problem that prevents the subject from completing required follow up.
21. Patient had a subarachnoid haemorrhage within 1 month prior to enrolment date.
22. Patient has a non-treated arterio-venous malformation in the territory of the target aneurysm.
23. Patient has a need for long-term use of anticoagulants.
24. Patient who is unable to complete the required follow-up.
25. Inability to understand the study or history of non-compliance with medical advice.
26. Evidence of active infection at the time of treatment.
27. Patient who is pregnant or breastfeeding.
28. Patient who has participated in a drug study within the last 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events following the eCLIPs procedure | Within 30 days of the procedure
  Proportion of subjects experiencing a device-related serious adverse event within 30 days following the procedure

SECONDARY OUTCOMES:
Technical Success | During Procedure
  Proportion of subjects with procedural success for the Electrolytic eCLIPs Bifurcation System. Procedural success defined as: access to the aneurysm, successful deployment, implantation of the eCLIPs Implant, and successful neck bridging of the target aneurysm, as judged by core lab evaluation of the procedural angiogram.
Success of adjuvant coiling | During Procedure
  Proportion of subjects with procedural success for the ability to insert coils into the aneurysm beyond the successfully implanted eCLIPs Implant, and the eCLIPs Implant to satisfactorily retain coils; irrespective of coil density or degree of occlusion.
Aneurysm Occlusion | At 6 month and 12 month follow-up
  Proportion of subjects with successful aneurysm treatment with the eCLIPs Implant and embolic coils, as measured by aneurysm occlusion of Modified Raymond-Roy Classification of 1 (no aneurysmal opacification) or 2 (residual neck) using DSA
Major ipsilateral stroke or neurologic death | Within12 months of procedure
  Proportion of subjects experiencing major stroke of neurologic death within 30 days, 6 and 12 months following the procedure.
All device-related adverse events (AEs) | Within 12 months of procedure
  A quantitative and descriptive summary of all device-related AEs experienced within 30 days, 6 and 12 months following the procedure.
Deterioration in modified Rankin Scale (mRS) score at Follow up | 30 days, 6, and 12 months following the procedure
  Proportion of subjects experiencing deterioration of modified Rankin Scale (mRS) score from baseline to 30 days, 6 and 12 month follow-up. Neurologic evaluation must be performed by independent qualified personnel.
Assessment of implant migration | 6 and 12 months following procedure
  Proportion of subjects with implant migration at 6 and 12 months follow up. Migration is defined as movement of the eCLIPs implant by 5mm compared to the position at implantation per core lab evaluation.
Assessment of branch artery patency | 6 and 12 months following procedure
  Proportion of subjects whose branch arteries (of the target aneurysm) are patent at 6 and 12 month follow up per core lab evaluation.
Patient Outcomes - Hospitalization length of stay (LOS) | Within 12 months of procedure
  Mean hospitalization LOS for index procedure.
Patient Outcomes - Subsequent hospitalization | Within 12 months of procedure
  Proportion of subjects requiring any subsequent hospitalization related to the index aneurysm.
Patient Outcomes - Remedial actions required | Within 12 months of procedure
  Proportion of subjects requiring remedial action for an adverse event during index procedure.
Patient Outcomes - Reintervention required | 30 days, 6, and 12 months following the procedure
  Proportion of subjects with complications, neurologic deterioration or adverse events requiring reintervention.
Patient Outcomes - Return to baseline or improved functioning | 6 and 12 months following procedure
  Proportion of subjects returning to baseline functioning or improved functioning as measured by modified Rankin Scale (mRS). Baseline mRS compared to mRS at follow up.
Patient Outcomes - Aneurysm recurrence | Within 30 days, 6, and 12 months following the procedure
  Proportion of subjects with index aneurysm recurrence.
Patient Outcomes - Aneurysm rupture | Within 30 days, 6, and 12 months following the procedure
  Proportion of subjects with index aneurysm rupture.
Patient Outcomes - Neurologic deterioration | Immediate post-procedure prior to discharge
  Proportion of subjects with neurologic deterioration pre-discharge.

IPD SHARING:
Plan to Share IPD: No